CLINICAL TRIAL: NCT01309698
Title: An Open-label, Randomized and Crossover Study to Assess the Effect of Co-administration of Vildagliptin and Voglibose on the Steady-state Pharmacokinetics / Pharmacodynamics in Japanese Patients With Type 2 Diabetes
Brief Title: Drug Interaction of Vildagliptin (LAF237) With Voglibose in Japanese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CLAF237A1103
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-11

CONDITIONS: Type 2 Diabetes
Keywords: Drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine; voglibose

ARMS (6):
- Treatment Sequence 1 (Experimental)
  Interventions: Drug: Vildagliptin (LAF237); Drug: Voglibose; Drug: Vildagliptin and Voglibose
- Treatment Sequence 2 (Experimental)
  Interventions: Drug: Vildagliptin (LAF237); Drug: Voglibose; Drug: Vildagliptin and Voglibose
- Treatment Sequence 3 (Experimental)
  Interventions: Drug: Vildagliptin (LAF237); Drug: Voglibose; Drug: Vildagliptin and Voglibose
- Treatment Sequence 4 (Experimental)
  Interventions: Drug: Vildagliptin (LAF237); Drug: Voglibose; Drug: Vildagliptin and Voglibose
- Treatment Sequence 5 (Experimental)
  Interventions: Drug: Vildagliptin (LAF237); Drug: Voglibose; Drug: Vildagliptin and Voglibose
- Treatment Sequence 6 (Experimental)
  Interventions: Drug: Vildagliptin (LAF237); Drug: Voglibose; Drug: Vildagliptin and Voglibose

INTERVENTIONS:
Drug: Vildagliptin (LAF237)
Drug: Voglibose
Drug: Vildagliptin and Voglibose

SUMMARY:
This study will evaluate the effect of voglibose on the pharmacokinetics and pharmacodynamics of vildagliptin in Japanese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with inadequately controlled on diet therapy and exercise therapy (HbA1c in the range 6.5 to 10.0% inclusive by NGSP)

Exclusion Criteria:

* Fasting plasma glucose ≥ 270 mg/dL A history of Type 1 diabetes or secondary forms of diabetes Treatment of anti-diabetic agents including GLP-1 analogues within 8 weeks or insulin within 6 months prior to screening Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of vildagliptin | Up to 12 hours post-dose

SECONDARY OUTCOMES:
Pharmacodynamic parameters (dipeptidyl peptidase IV (DPP-4) activity, glucagon-like peptide-1(GLP-1), glucose, insulin, glucagon) | Up to 4 hours or 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Tokyo, Japan

REFERENCES:
- [Result] Yamaguchi M, Saji T, Mita S, Kulmatycki K, He YL, Furihata K, Sekiguchi K. Pharmacokinetic and pharmacodynamic interaction of vildagliptin and voglibose in Japanese patients with Type 2 diabetes. Int J Clin Pharmacol Ther. 2013 Aug;51(8):641-51. doi: 10.5414/CP201902. PMID 23782587
- See also: Results for CLAF237A1103 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5843